CLINICAL TRIAL: NCT03931044
Title: Fluorescence Image-Guided Lymphadenectomy Using Indocyanine Green and Near Infrared Technology in Robotic Gastrectomy
Brief Title: Fluorescence Image-Guided Lymphadenectomy in Robotic Gastrectomy
Acronym: IG-MIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Study Group on Minimally Invasive Surgery for Gastric Cancer (Other)
Responsible Party: Principal Investigator, Amilcare Parisi, Director of the Department of Digestive Surgery - St. Mary's Hospital of Terni, International Study Group on Minimally Invasive Surgery for Gastric Cancer
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IG-MIG Vers. 1.0-05.03.2019
Record Dates: First submitted 2019-04-21; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Gastric Cancer; Sentinel Lymph Node
Keywords: Robotic surgery; fluorescence; indocyanine green; lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image-Guided Robotic Gastrectomy (Experimental): The day before surgery, the ICG will be injected endoscopically into the submucosa of the four quadrants around the tumor (1.25mg/mL, 0.6mL x 4).
  A modified total D2 gastrectomy - including the following lymph node stations: 1 - 7 + 8a, 9, 11p, 12a - will be performed in each patient.
  The lymph node dissection will be performed using the Da Vinci Xi robotic system and the assistance of the near infrared technology to detect ICG fluorescence.
  Even the resulting fluorescent lymph nodes outside the standard dissection plane will be retrieved. The lymph node stations will be sent to the pathologist in different containers and further subdivided according to fluorescence.
  Interventions: Procedure: Image-Guided Robotic Gastrectomy
- Robotic Gastrectomy (No Intervention): Data from patients undergoing the same surgery without the ICG imaging procedure will be collected during the same study period.

INTERVENTIONS:
Procedure: Image-Guided Robotic Gastrectomy — The near-infrared technology, integrated in the robotic camera, will be used to detect fluorescent lymphonodes.
  Arms: Image-Guided Robotic Gastrectomy

SUMMARY:
Gastric cancer is a worldwide challenge due to its spread, even epidemic in some areas, and the high mortality rates. Lymphadenectomy is considered the fundamental step during radical gastrectomy. In recent years, some researchers have tried to find a way to improve the surgical identification of the lymphatic drainage routes and lymph node stations. This new surgical frontier is the so called "navigation surgery". Among the different reported solutions, lately, the indocyanine green (ICG) has drawn attention. It is a fluorescence dye, that can be detected in the near infrared spectral band (NIR). The development of specific fluorescence imaging devices has allowed surgeons to visualize tumors, vascular and lymphatic structures. The Da Vinci Xi robotic system has an integrated imaging technology that has been used in colo-rectal and hepato-biliary surgery. However, up to date, the combined use of fluorescence imaging and robotic technology has not been evaluated during lymphadenectomy in gastric cancer.

The general design of the present study is to evaluate the role of fluorescence imaging during robotic lymphadenectomy for gastric cancer.

DETAILED DESCRIPTION:
Background Gastric cancer is the fourth most widespread cancer in the world and is characterized by high mortality rates [1, 2]. A multidisciplinary context, in which surgery plays the main role, is essential to offer the best therapeutic strategy. Lymph node involvement in gastric cancer is present in 2-18% when the depth of the tumor invasion is limited to the mucosal or submucosal layer, but rises to 50% when the tumor involves the subserosa [3]. Lymphadenectomy is a fundamental surgical phase that must guarantee the oncological radicality and allow an appropriate tumor staging. Although it is among the most relevant factors influencing long-term survival, its extension and standardization is still the subject of much debate. The two latest editions of the Japanese Gastric Cancer Association (JGCA) guidelines [4] recommend a dissection on different levels (D1, D1 +, D2) depending on the type of gastrectomy and the clinical stage of the tumor. In recent years, some researchers have tried to apply the concept of "sentinel lymph node" to gastric cancer [5-7]. Although some do not consider that terminology the appropriate one in the context of gastric cancer, because of the multidirectional gastric lymphatic flows, several studies have highlighted interesting aspects, such as: limiting an extensive lymphatic dissection when not necessary, identifying the drainage routes outside the standard anatomical planes, possible assistance in minimally invasive procedures [8]. Most of the experiences in lymph nodes mapping were performed with a radio-isotope (Tc99m) associated or not with the intraoperative use of vital dyes (Blue dye). More recently, the properties of the ICG have been studied. This is a fluorescence dye, that can be detected in the NIR [9, 10]. The development of imaging tools using "NIR / ICG" technology is therefore an innovative approach for visualizing tumors, vascular structures, lymphatic channels, and lymph nodes [11]. Some advantages of the ICG are: reduced toxicity, absence of radioactivity, low cost, safe administration both intravenously and endoscopically through the submucosa or subserosa, protein binding without changing molecular structures, macrophages interaction at the lymph node level. Devices for fluorescence imaging are currently available in both open and minimally invasive surgery.

In this field, robotic surgery has been becoming of great interest thanks to the manufacturing of new instruments which, compared to laparoscopy, allow to improve manual skills and gentleness in challenging movements [12]. The Da Vinci Xi robotic system has also produced an innovative imaging technology for ICG visualization made up with a laser source integrated in the robotic camera (Firefly). The surgeon at the console has therefore a 3-D vision that can switch to the fluorescence mode without the need to change the camera. Few clinical experiences have been reported to date [12]. Published articles refer to assistance in colo-rectal and hepato-biliary surgery for vessels or biliary structures visualization, while its use during lymph node dissection for gastric cancer has not yet been the subject of study protocols.

Hypothesis: fluorescence imaging during lymphadenectomy in gastric cancer can significantly improve the quality of the dissection through a better visualization of anatomical planes and allow tailored dissections. Moreover, the tumor status in the fluorescent nodes could predict the nodes status in the overall specimen with high accuracy rate.

Methods General study design: the overall objective is verifying the feasibility and the role of a lymphadenectomy assisted by fluorescence imaging during robotic gastrectomy.

Two levels of investigation are planned:

* to detect the possible advantages of a fluorescence-guided surgery ("Navigation Surgery");
* to evaluate the possibility of considering the lymph nodes labeled by the ICG as predictive of the state of tumor diffusion ("Targeted Surgery") Type of study: Interventional study.

Specific aims:

1. To verify the ability of the procedure to highlight the main tumor lymphatic drainage pathways.
2. To validate the concept of Navigation Surgery in gastric surgery by comparing the group of the experimental procedure with a control group undergoing the same type of surgery but not assisted by fluorescence.
3. To find a correlation between the nodes marked by the ICG and the remaining nodes removed during the procedure.
4. To identify the characteristics of those patients in whom the ICG can effectively discriminate the type of lymphadenectomy to be performed.

Data collection: the following information will be collected for each patient.

- General variables: demographic, histopathological, intra and post-operative features, complications. - Specific variables: total number of lymph nodes retrieved (LNs), Fluorescent lymph nodes (FLNs), metastatic LNs, LNs by station, FLNs outside the standard dissection plane, FLNs status (positive or negative for tumor), non-fluorescent LNs status

Definitions and subdivision of patients:

* True positive patients: patients in which FLNs positive for tumor are detected when LNs positive for tumor are found in the analysis of the surgical specimen.
* False positive patients: patients in which FLNs positive for tumor are detected when LNs negative for tumor are found in the analysis of the surgical specimen.
* True negative patients: patients in which FLNs negative for tumor are detected when LNs negative for tumor are found in the analysis of the surgical specimen.
* False negative patients: patients in which FLNs negative for tumor are detected when LNs positive for tumor are found in the analysis of the surgical specimen.

Sample size: considering the volume of patients included in published studies available in the literature on the use of fluorescence imaging and adding that the present project is the first to describe the use of robotic technology with fluorescence assistance in gastric cancer, a total of 20 patients will be enrolled for the experimental procedure. An additional sample including 20 patients will be the control group, based on the same eligibility criteria. The total sample of patients planned for the present study is therefore of 40 subjects.

Statistical analysis: SPSS v23 will be used to perform data analysis. The dichotomous variables will be expressed as numbers and percentages, while the continuous variables as mean and standard deviation, or median and IQR (minimum and maximum values). For the comparison with the control group, the continuous variables will be analyzed with the T test for independent samples and a value of P <0.05 will be considered statistically significant.

Impact on clinical practice and healthcare system: this project can pave the way for a new concept of lymphadenectomy in gastric cancer involving minimally invasive surgery. Patients could benefit from a more tailored approach to their disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of gastric cancer proved through the endoscopic biopsy
* cT1 - cT3
* cN0

Exclusion Criteria:

* history of allergies related to iodine
* pregnancy
* cT4,
* cN +
* distant metastases
* estimated sizes > 4cm
* synchronous malignant tumors in other organs
* ASA score ≥ 4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mean difference of total number of LNs retrieved during surgery (mean±DS) | 1 year
  Usefulness of the Navigation Surgery through a comparison between the two groups on the number of LNs retrieved
FLNs identification rate (No, %) | 1 year
  Patients in which the procedure detects FLNs.
Accuracy (%; 95% CI) | 1 year
  Degree of deviation between the FLNs tumor status and the status found in the other LNs analyzed. [true positive patients + true negative patients / TOT patients]

SECONDARY OUTCOMES:
Mean difference of total number of LNs retrieved during the lymphadenectomy of the D2 anatomical plane (mean±DS). | 1 year
  Impact on the D2 lymph node dissection through a comparison between the two groups on the number of LNs removed in the D2 anatomical plane.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale di Forlì "G.B. Morgagni" - AUSL della Romagna - U.O.C. di Chirurgia e Terapie Oncologiche Avanzate, Forlì
  - Azienda Ospedaliera di Terni "Santa Maria" - S.C. di Chirurgia Digestiva, Terni

REFERENCES:
- [Background] Bray F, Jemal A, Grey N, Ferlay J, Forman D. Global cancer transitions according to the Human Development Index (2008-2030): a population-based study. Lancet Oncol. 2012 Aug;13(8):790-801. doi: 10.1016/S1470-2045(12)70211-5. Epub 2012 Jun 1. PMID 22658655
- [Background] Hartgrink HH, Jansen EP, van Grieken NC, van de Velde CJ. Gastric cancer. Lancet. 2009 Aug 8;374(9688):477-90. doi: 10.1016/S0140-6736(09)60617-6. Epub 2009 Jul 20. PMID 19625077
- [Background] Sasako M, McCulloch P, Kinoshita T, Maruyama K. New method to evaluate the therapeutic value of lymph node dissection for gastric cancer. Br J Surg. 1995 Mar;82(3):346-51. doi: 10.1002/bjs.1800820321. PMID 7796005
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Kitagawa Y, Fujii H, Mukai M, Kubota T, Otani Y, Kitajima M. Radio-guided sentinel node detection for gastric cancer. Br J Surg. 2002 May;89(5):604-8. doi: 10.1046/j.1365-2168.2002.02065.x. PMID 11972551
- [Background] Kitagawa Y, Takeuchi H, Takagi Y, Natsugoe S, Terashima M, Murakami N, Fujimura T, Tsujimoto H, Hayashi H, Yoshimizu N, Takagane A, Mohri Y, Nabeshima K, Uenosono Y, Kinami S, Sakamoto J, Morita S, Aikou T, Miwa K, Kitajima M. Sentinel node mapping for gastric cancer: a prospective multicenter trial in Japan. J Clin Oncol. 2013 Oct 10;31(29):3704-10. doi: 10.1200/JCO.2013.50.3789. Epub 2013 Sep 9. PMID 24019550
- [Background] Kitagawa Y, Fujii H, Kumai K, Kubota T, Otani Y, Saikawa Y, Yoshida M, Kubo A, Kitajima M. Recent advances in sentinel node navigation for gastric cancer: a paradigm shift of surgical management. J Surg Oncol. 2005 Jun 1;90(3):147-51; discussion 151-2. doi: 10.1002/jso.20220. PMID 15895450
- [Background] Tani T, Sonoda H, Tani M. Sentinel lymph node navigation surgery for gastric cancer: Does it really benefit the patient? World J Gastroenterol. 2016 Mar 14;22(10):2894-9. doi: 10.3748/wjg.v22.i10.2894. PMID 26973385
- [Background] Vahrmeijer AL, Hutteman M, van der Vorst JR, van de Velde CJ, Frangioni JV. Image-guided cancer surgery using near-infrared fluorescence. Nat Rev Clin Oncol. 2013 Sep;10(9):507-18. doi: 10.1038/nrclinonc.2013.123. Epub 2013 Jul 23. PMID 23881033
- [Background] Yoshida M, Kubota K, Kuroda J, Ohta K, Nakamura T, Saito J, Kobayashi M, Sato T, Beck Y, Kitagawa Y, Kitajima M. Indocyanine green injection for detecting sentinel nodes using color fluorescence camera in the laparoscopy-assisted gastrectomy. J Gastroenterol Hepatol. 2012 Apr;27 Suppl 3:29-33. doi: 10.1111/j.1440-1746.2012.07067.x. PMID 22486868
- [Background] Bu L, Shen B, Cheng Z. Fluorescent imaging of cancerous tissues for targeted surgery. Adv Drug Deliv Rev. 2014 Sep 30;76:21-38. doi: 10.1016/j.addr.2014.07.008. Epub 2014 Jul 24. PMID 25064553
- [Background] Marano A, Priora F, Lenti LM, Ravazzoni F, Quarati R, Spinoglio G. Application of fluorescence in robotic general surgery: review of the literature and state of the art. World J Surg. 2013 Dec;37(12):2800-11. doi: 10.1007/s00268-013-2066-x. PMID 23645129